CLINICAL TRIAL: NCT00575692
Title: Magnetic Resonance Imaging in the Diagnosis of Pulmonary Hypertension
Status: Completed | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Principal Investigator, Olschewski, Horst, Prof. MD, Univ.-Prof. Dr., Medical University of Graz
Other Study IDs: PH-06-CMR-01
Record Dates: First submitted 2007-12-17; First posted 2007-12-18 (Estimated); Last update posted 2014-05-28 (Estimated); Status verified 2014-05

CONDITIONS: Pulmonary Hypertension; Ventricular Function; MR Phase Contrast Velocity Imaging; Late Enhancement Patterns
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- PulmoHypertension: Patients with suspected, latent or manifest pulmonary hypertension
- Controls: Controls without history of cardiac or pulmonary diseases

SUMMARY:
The aim of the present study is to identify changes in the cardiovascular system in patients with pulmonary hypertension (PH) by magnetic resonance imaging (MRI). MRI is accepted as golden standard method for the evaluation of left and right ventricular morphology and function.

All patients who showed elevated pulmonary pressure in the right heart catheter investigation are assigned to MRI. Parameters derived from MRI are included in the clinical and therapeutic decisions. Well established as well as new MRI parameters are evaluated and compared to the results of right heart catheter. Further age-matched controls without known cardiac or pulmonary disease are investigated by native MRI.

DETAILED DESCRIPTION:
Patients with suspected, latent and manifest PH and controls are investigated by MRI according to the following protocol in breathhold or free breathing (depending on the patients' breath-hold abilities). In case of elevated Creatinin values, no contrast agent is applied.

* Planning of cardiac views: Planning of 2-chamber view, short axes view and 4-chamber view.
* Morphological overview: Transversal and coronal Haste images
* Left and right heart functional and valve evaluation: Cine 2-chamber imaging, Multi-slice cine 4-chamber imaging, Cine Left and Right ventricular outflow tract imaging and Multi-slice cine short axes imaging covering the left and right ventricle for evaluation of EDV, ESV, SV, EF, CO and muscle mass.
* Phase Contrast Imaging: Flow measurements in the aorta, the pulmonary artery and the heart.
* Perfusion measurement.
* Late enhancement measurement: Multi-slice short axes view, multi-slice 2-chamber view and multi-slice 4-chamber view.

ELIGIBILITY:
Inclusion Criteria:

* Controls without history of cardiac or pulmonary diseases
* Patients with suspected PH
* Patients with latent PH
* Patients with manifest PH

Exclusion Criteria:

* MRI exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cardiac MR is recommended to all patients with suspected, latent and manifest PH who are investigated by right heat catheter in the Department of Pulmonology. Patients with pacemaker, agoraphobia or other standard MR contraindications are excluded from the study.
Sampling Method: Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2006-12; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
right ventricular function | at the MRI investigation
  right ventricular end-diastolic volume (EDV), right ventricular end-systolic volume (ESV), right ventricular stroke volume (SV), right ventricular ejection fraction (EF), right ventricular cardiac output (CO), right ventricular muscle mass (RVMM)

CONTACTS AND LOCATIONS:
Overall Officials: Gabor Kovacs, MD, Principal Investigator — Medical Unitersity Graz, University Clinic of Internal Medicine, Department of Pulmonology; Ursula Reiter, PhD, Principal Investigator — Medical Unitersity Graz, University Clinic of Radiology, Department of General Radiological Diagnostics; Gert Reiter, PhD, Principal Investigator — Siemens Medical Austria; HOrst Olschewski, M.D., Principal Investigator — Medical University of Graz
Locations (1):
- Medical Unitersity Graz, University Clinic of Internal Medicine, Department of Pulmonology, Graz, Stmk., Austria

REFERENCES:
- [Result] Reiter G, Reiter U, Kovacs G, Kainz B, Schmidt K, Maier R, Olschewski H, Rienmueller R. Magnetic resonance-derived 3-dimensional blood flow patterns in the main pulmonary artery as a marker of pulmonary hypertension and a measure of elevated mean pulmonary arterial pressure. Circ Cardiovasc Imaging. 2008 Jul;1(1):23-30. doi: 10.1161/CIRCIMAGING.108.780247. PMID 19808511
- [Derived] Reiter G, Kovacs G, Reiter C, Schmidt A, Fuchsjager M, Olschewski H, Reiter U. Left atrial acceleration factor as a magnetic resonance 4D flow measure of mean pulmonary artery wedge pressure in pulmonary hypertension. Front Cardiovasc Med. 2022 Aug 3;9:972142. doi: 10.3389/fcvm.2022.972142. eCollection 2022. PMID 35990987
- [Derived] Reiter U, Kovacs G, Reiter C, Krauter C, Nizhnikava V, Fuchsjager M, Olschewski H, Reiter G. MR 4D flow-based mean pulmonary arterial pressure tracking in pulmonary hypertension. Eur Radiol. 2021 Apr;31(4):1883-1893. doi: 10.1007/s00330-020-07287-6. Epub 2020 Sep 24. PMID 32974687
- [Derived] Reiter G, Reiter U, Kovacs G, Olschewski H, Fuchsjager M. Blood flow vortices along the main pulmonary artery measured with MR imaging for diagnosis of pulmonary hypertension. Radiology. 2015 Apr;275(1):71-9. doi: 10.1148/radiol.14140849. Epub 2014 Nov 5. PMID 25372980